CLINICAL TRIAL: NCT00826397
Title: Pilot Study on the Effect of Acupuncture on Joint Pain Induced by Aromatase Inhibitors in Breast Cancer Patients
Brief Title: Acupuncture for Aromatase Inhibitor Induced Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Dawn L. Hershman, Associate Professor of Medicine & Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AAAB2299
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
Keywords: Aromatase Inhibitors; Joint Pain; Symptoms Control; Acupuncture
MeSH Terms: conditions — Breast Neoplasms; Arthralgia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Arm (Experimental): Patients in the treatment arm will receive acupuncture administered twice weekly for six weeks and will be allowed to take pain medication as necessary.
  Interventions: Procedure: Acupuncture
- Control Arm (Sham Comparator): The control patients will receive a form of sham acupuncture, which will consist of superficial needling at nonspecific body points, administered twice weekly for six weeks.
  Interventions: Procedure: Sham Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Each acupuncture session will last approximately 45 minutes and includes standardized body treatment with an emphasis on affected joints.
  Arms: Acupuncture Arm
Procedure: Sham Acupuncture — The sham acupuncture session will consist of superficial needling at nonspecific body points, administered twice weekly for six weeks, and will last approximately 45 minutes and includes standardized body treatment with an emphasis on affected joints.
  Arms: Control Arm

SUMMARY:
This is a randomized, controlled, pilot study to determine the safety and efficacy of acupuncture as an adjunct to pharmacological treatment compared to pharmacological intervention alone for the treatment of musculoskeletal pain related to aromatase inhibitors (AI) in postmenopausal breast cancer patients. Twenty participants (20 in each arm) will be enrolled at the Breast Oncology clinic at Columbia University Medical Center (CUMC). Patients in the treatment arm will receive acupuncture administered twice weekly for six weeks and will be allowed to take pain medication as necessary. The control patients will initially receive pain medication alone, then will cross-over to the acupuncture arm after six weeks. The investigators hypothesize that acupuncture will reduce AI induced joint symptoms.

The study will enroll a total of 40 patients, half of whom will be randomized to one of the two arms to receive acupuncture plus pharmacological treatment (arm A) or pharmacological treatment alone (arm B). Joint pain will be assessed by the BPI-SF score at baseline and six weeks. All patients will have a baseline BPI worst pain item (#2) ≥3 points on a scale of 0-10.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and efficacy of acupuncture as a complementary therapy to pain medication for joint pain associated with aromatase inhibitors for breast cancer treatment. Breast cancer patients are living longer largely due to the benefits of hormonal therapy. Aromatase inhibitors (AIs) are a new class of hormonal agents which block estrogen synthesis in postmenopausal women. However, musculoskeletal pain occurs in up to 50% of patients treated with AIs and often does not respond to conventional pain medications. AI-induced joint pain interferes with patient compliance and may cause major disability. Therefore, safe and effective treatments are needed to alleviate AI-induced musculoskeletal pain.

Acupuncture is a traditional Chinese method of medical treatment and a popular modality for treating musculoskeletal pain. Acupuncture involves the use of thin needles to stimulate specific points of the body and leads to pain control through the release of endorphin in the central nervous system. Clinical trials have found a benefit of acupuncture for the treatment of knee and back pain. Given the lack of effective treatments for AI-induced joint pain and the safety and efficacy of acupuncture, it is therefore reasonable to evaluate whether acupuncture is effective in breast cancer patients who experience musculoskeletal pain related to AIs.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age>45 years
* Postmenopausal status defined as cessation of menses for >1 year or follicle- stimulating hormone (FSH)>20 mIU/mL
* History of stage I or II, hormone receptor-positive breast cancer
* Currently taking a third-generation aromatase inhibitor (anastrazole, letrozole or exemestane)
* Ongoing musculoskeletal pain in one or more joints (baseline BPI worst pain score > 3 points on a scale of 0 to 10)
* English-speaking
* Signed informed consent

EXCLUSION CRITERIA:

* Previous treatment with acupuncture
* Inflammatory, metabolic or neuropathic arthropathies
* Bone fracture or surgery of the afflicted extremity during the past six months
* Current narcotic use, corticosteroid therapy or cortisone injections
* Severe concomitant illnesses or metastatic disease
* Severe coagulopathy or bleeding disorder
* Dermatological disease within the acupuncture area

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in Joint Pain | Baseline and 6 weeks
  This is defined as the difference in the Brief Pain Inventory - Short Form (BPI-SF) scale at six weeks versus baseline.

SECONDARY OUTCOMES:
Change in Joint Stiffness and Function | Baseline and 6 weeks
  The Western Ontario and McMaster Universities Osteoarthritis (WOMAC) index Version 3.1 will be used and consists of 24 questions related to three subscales: pain (0-20), stiffness (0-8) and physical function (0-68).
Safety and Tolerability measured by Frequency of Adverse Events | 6 weeks
  Reporting of the severity and frequency of adverse events (NCI Common Terminology Criteria Version 3.0) (40) related to the interventions will be conducted every two weeks during telephone interviews. All treatment-related adverse events will be reported for both treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided